CLINICAL TRIAL: NCT01150656
Title: SCOR in Targeted Therapies for Infant Leukemias Project 2: Targeting Apoptosis in Leukemia in Infants
Brief Title: Obatoclax Mesylate in Samples From Young Patients With Acute Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AAML10B17; COG-AAML10B17 (Other: Children's Oncology Group); NCI-2011-02239 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AAML10B17 (Other: Children's Oncology Group)
Record Dates: First submitted 2010-06-24; First posted 2010-06-25 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Leukemia
Keywords: childhood acute myeloid leukemia/other myeloid malignancies
MeSH Terms: conditions — Leukemia | interventions — Gene Expression Profiling; Microarray Analysis; Reverse Transcriptase Polymerase Chain Reaction; Blotting, Western

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: gene expression analysis
Genetic: microarray analysis
Genetic: protein expression analysis
Genetic: reverse transcriptase-polymerase chain reaction
Genetic: western blotting
Other: laboratory biomarker analysis
Other: pharmacological study

SUMMARY:
RATIONALE: Studying the effects of obatoclax mesylate in cell samples from patients with cancer in the laboratory may help doctors learn more about the effects of obatoclax mesylate on cancer cells. It may also help doctors identify biomarkers related to cancer.

PURPOSE: This research study is studying obatoclax mesylate in samples from young patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine comprehensive gene and protein expression profiles of in vitro sensitivity and resistance to obatoclax mesylate in multiple-lineage leukemia (MLL)-rearranged cell lines and primary infant acute myeloid leukemia (AML) samples.
* Define optimum in vitro combinations of obatoclax mesylate targeting pro-survival BCL-2 family proteins with cytotoxic drugs in MLL-rearranged leukemia cell lines and primary infant AML samples.
* Identify synergistic combinations based on a pharmacodynamic modeling and simulation construct.
* Determine whether combinations of obatoclax mesylate targeting pro-survival BCL-2 family proteins with cytotoxic drugs improves survival in a xenograft model of MLL-rearranged infant AML.

OUTLINE: This is a multicenter study.

Obatoclax mesylate activity is assessed via the MTT assay. A priori features of acute myeloid leukemia (AML) blasts relating to the apoptosis and ATG cell death pathways and their execution are characterized using microarray analysis and quantitative real-time (Q-RT) PCR. Gene and protein expression is described and quantified using Q-RT PCR and western blot analysis at specific time points after obatoclax mesylate exposure to identify pharmacodynamic biomarkers of activity and characterize the cell death mechanism in multiple-lineage leukemia (MLL)+ AML. The MTT assay is performed using obatoclax mesylate-cytotoxic chemotherapy combinations to determine synergy focusing on common cytotoxic drugs employed in AML treatment regimens.

Obatoclax mesylate efficacy is tested in a therapeutic NOG xenograft model of primary MLL+ infant AML.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute myeloid leukemia (AML)
* Cryopreserved samples from infants with AML available

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients With Acute Myeloid Leukemia
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2010-06; Primary Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Obatoclax mesylate activity
Optimum in vitro combinations of obatoclax mesylate
Pharmacodynamic (PD) biomarkers of activity
Cell death mechanism in multiple-lineage leukemia (MLL) acute myeloid leukemia (AML)
Disease progression in a xenograft model of MLL-rearranged infant AML

SECONDARY OUTCOMES:
Physical assessment (in xenograft model)
Peripheral blast count reduction
Apoptosis and/or ATG induction
Modulation of relevant PD biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn A. Felix, MD, Principal Investigator — Children's Hospital of Philadelphia